CLINICAL TRIAL: NCT04937972
Title: SHR-1701 Combined With Fluzoparib as Maintenance Therapy for Advanced Lung Squamous Cell Carcinoma After Platium Based Chemo-immunotherapy
Brief Title: SHR-1701 Combined With Fluzoparib in Lung Squamous Cell Carcinoma
Acronym: FLYFLY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, HunanPTH, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701
Record Dates: First submitted 2021-06-18; First posted 2021-06-24 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701 Combined With fluzoparib (Experimental)
  Interventions: Drug: SHR-1701 Combined With Fluazopalil

INTERVENTIONS:
Drug: SHR-1701 Combined With Fluazopalil — SHR-1701 +fluzoparib

SUMMARY:
The purpose of the trial was to evaluate the efficacy and safety of SHR-1701 combined with fluzopar as a first-line treatment maintenance therapy for advanced lung squamous cell carcinoma. Patients with advanced or metastatic (stage IV) lung squamous cell carcinoma have not received systemic chemotherapy and have measurable lesions (RECIST 1.1) ECOG PS 0-1. The patient received SHR1701 +fluzoparib

ELIGIBILITY:
Inclusion Criteria:

* 1.The age at the time of signing the informed consent form is 18-75 years old, both male and female;
* 2.Advanced or metastatic lung squamous cell carcinoma confirmed by histology or cytology;
* 3.Has not received systemic treatment for the recurrence or metastasis stage in the past. If you have received neoadjuvant or adjuvant chemotherapy/radiotherapy in the past, those who have relapsed or metastasized> 6 months from the end of treatment can be included in the group.
* 4.ECOG PS score: 0-1 points;
* 5.According to the RECIST 1.1 standard, the patient must have at least one measurable lesion;
* 6.The function of major organs is normal, that is, it meets the following standards: a) Routine blood examination (under 14 days without blood transfusion and no hematopoietic stimulating factor drugs for correction): hemoglobin (Hb) ≥90g/L; absolute neutrophil count (ANC) ) ≥1.5×109/L; platelet (PLT) ≥100×109/L; white blood cell count (WBC) ≥3.0×109/L; b) Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ×Upper limit of normal (ULN); serum total bilirubin (TBIL)≤1.5×ULN; serum creatinine (Cr)≤1.5×ULN or creatinine clearance ≥50ml/min; c) coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT)≤1.5×ULN; d) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF)≥50%;
* 7.Expected survival period ≥ 3 months; Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug; for men, surgical sterilization should be performed Or agree to use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug;
* 8.The patient voluntarily participates and signs the informed consent form (or signed by the legal representative). It is expected to have good compliance and be able to cooperate with the research according to the requirements of the plan.

Exclusion Criteria:

* 1) Untreated brain metastases (persons who have previously received treatment for brain metastases (radiotherapy or surgery), if the images have been confirmed to be stable for at least 4 weeks before randomization, and systemic hormone therapy has been discontinued (dose>10mg/day prednisone or Other equivalent hormones), those without clinical symptoms can be included in the group);
* 2) With meningeal metastasis, spinal cord compression, etc.;
* 3) Patients with pleural effusion, pericardial effusion or ascites who need to be drained with clinical symptoms, or who have received drainage of serous cavity effusion for treatment purposes within 2 weeks before randomization;
* 4) Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] test results are positive, HBV-DNA ≥ 500 IU/ml and abnormal liver function; hepatitis C is defined as hepatitis C antibody [HCV-Ab] positive, HCV-RNA higher than the detection limit of the analysis method and abnormal liver function) or combined hepatitis B and C co-infection ；
* 5) Suffer from any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (hormone replacement) Can be included after treatment)); patients with childhood asthma have been completely relieved and no intervention is required after adulthood or vitiligo can be included, and patients who require medical intervention with bronchodilators cannot be included;
* 6) Severe infection (such as intravenous infusion of antibiotics, antifungal or antiviral drugs required) within 2 weeks before the first administration, or unexplained fever >38.5°C during the screening period/before the first administration;
* 7) Arterial/venous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
* 8) Persons with a history of significant clinical significance of cardiovascular disease, including but not limited to; (1) Congestive heart failure (NYHA grade> 2); (2) Unstable angina pectoris; (3) 3 months before signing the ICF Myocardial infarction occurred within; (4) Any supraventricular arrhythmia or ventricular arrhythmia that requires treatment or intervention;
* 9) Suffered from or accompanied with other systemic malignancies in the last 5 years, (except for cured skin basal cell carcinoma, cervical carcinoma in situ and ovarian cancer);
* 10) Have received a preventive vaccine or attenuated vaccine within 4 weeks before the first administration;
* 11) Those who are known to be allergic to any test drug or its excipients;
* 12) Pregnant and lactating patients, and reproductive patients are unwilling to take effective contraceptive measures;
* 13) Have a clear history of neurological or mental disorders, including epilepsy and dementia;
* 14) Patients who are unable to swallow the study drug, such as chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis) and intestinal obstruction and other factors that affect drug intake and absorption;
* 15) Other situations that the researcher thinks are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)

SECONDARY OUTCOMES:
ORR | 1 year
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects
DCR | 1 year
  Defined as the proportion of subjects with complete remission (CR), partial remission (PR) and stable disease (SD) to the total subjects

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China